CLINICAL TRIAL: NCT03904121
Title: Colon Cancer Surgery in the Aged; Postoperative Outcome, Functional Recovery and Survival
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Susanna Niemeläinen, Chief Physician of Surgery, Tampere University Hospital
Other Study IDs: R19028
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Colon Cancer
Keywords: Colon cancer surgery octogenarian postoperative outcome
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Curative operation — Postoperative morbidity, mortality, functional outcome, survival
  Other Names: Palliative operation; Non-operative treatment

SUMMARY:
Patients aged > 80 years represent an increasing proportion of colon cancer diagnoses. It is important to have relevant and trustable data concerning elderly colorectal cancer patients surgery and postoperative morbidity, functional ability, life quality and survival numbers. With possibly compromised health status and functional decline the benefits of surgical management and outcomes can diminish life quality and overall survival.

With proper patients selection, preoperative health evaluation and thus patient information, colorectal cancer surgery can be performed with lower morbidity and mortality rates with comparative survival numbers.

The aim of this prospectively collected, observational study is to acquire data from colorectal cancer surgery in aged over 80 years and perform statistical analysis of the preoperative risk factors affecting postoperative morbidity, functional recovery, mortality and overall survival.

DETAILED DESCRIPTION:
9 Finnish hospitals including three university hospitals participate in the study. The data is collected from the hospitals using a specially designed and secure web application (RedCap).

The preoperative patients' data include comorbidities, clinical frailty scale (CFS) and functional status, postoperative surgical and medical outcomes and survival data. The patient questionnaire is based on the G-8 geriatric screening tool and MNA-short form. The questionnaire is filled out preoperatively and 1, 3, 6 and 12 months postoperatively. The patient data concerning procedures is collected from the hospitals prospectively recording data. Mortality data on causes of death are obtained from Statistics Finland.

All colon cancer patients aged over 80 years with curative disease (stage I-III) are included. Patients with metastatic disease or severe Alzheimer disease are excluded. They are treated either non-operatively or with curative resection or palliative procedure. Patients fill out the approval form. The study is acknowledged by the ethics committee of the participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* primary colon cancer, which is surgically treated with curative intent (stage I-III)

Exclusion Criteria:

* metastatic colon cancer, severe dementia, life expectancy less than six months

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary colon cancer patients (stage I-III) in the aged over 80 years
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity | 30 days
  Clavien-Dindo classification (0-V)
Postoperative mortality | 12 months
  Date of death

SECONDARY OUTCOMES:
Functional performance | 12 months
  Patient questionnaire ( nutritional status, mobility, use of implements, medication, weight, housing, homeaid), scale 0-3; 0= no, 1= sometimes, 2= often, 3= always

CONTACTS AND LOCATIONS:
Overall Officials: Marja Hyöty, M.D.,Ph.D., Study Director — Tampere UH
Locations (1):
- Tampere University, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niemelainen S, Huhtala H, Ehrlich A, Kossi J, Jamsen E, Hyoty M. Surgical and functional outcomes and survival following Colon Cancer surgery in the aged: a study protocol for a prospective, observational multicentre study. BMC Cancer. 2021 Jun 14;21(1):698. doi: 10.1186/s12885-021-08454-8. PMID 34126949